CLINICAL TRIAL: NCT04674410
Title: Utility of Empiric Antibiotics on Admission for Non-intubated Patients With Novel Coronavirus Diseases 2019 (COVID-19): A Retrospective Cohort Study of Electronic Health Records
Brief Title: Utility of Empiric Antibiotics for Non-intubated Novel Coronavirus Diseases 2019 Patients
Status: Withdrawn | Type: Observational
Why Stopped: Reduced relevance given end of pandemic
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Sameer Kadri, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Other Study IDs: BD022383
Record Dates: First submitted 2020-12-17; First posted 2020-12-19 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Covid19; Coronavirus Infection; Pneumonia
Keywords: Empiric antibiotics
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Pneumonia | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Empiric Antibiotic: All patients with COVID19 diagnosed on admission who received empiric antibiotics within 48 hours of admission without another site of infection identified or suspected septic shock.
  Interventions: Drug: Antibiotic
- Control group: All patients admitted with COVID19 who did not receive empiric antibiotics in the first 48 hours of admission

INTERVENTIONS:
Drug: Antibiotic — Empiric antibiotic therapy, subdivided according to Community Acquired Pneumonia coverage vs Hospital Acquired Pneumonia coverage
  Groups: Empiric Antibiotic

SUMMARY:
This retrospective analysis of inpatient data obtained from administrative and electronic medical records will investigate the role of empiric antibiotics on admission on the mortality for non-intubated patients presenting with Novel Coronavirus Diseases 2019 (COVID-19) associated pneumonia without extra-pulmonary sources of infection or septic shock.

DETAILED DESCRIPTION:
This study will examine the impact of empiric antibiotic therapy on patients who present to hospital with an acute lower respiratory illness and a diagnosis of COVID-19 present-on-admission.

The Premier Healthcare Database will be used as the data source for administrative data. In addition, the subset of hospitals reporting microbiology and laboratory data will be used for subset analyses and validation purposes. The primary population to be studied will be non-intubated patients diagnosed with COVID-19 on admission (identified by diagnosis coding and/or polymerase chain reaction result present-on-admission) who have diagnosis codes supportive of acute lung illness (e.g. pneumonia). Patients with extra-pulmonary infections present-on-admission for which antibiotics would be generally administered and/or those requiring vasopressors and/or mechanical ventilation on the day of admission or day after will be excluded.

Patients will be analyzed according to their antibiotic treatment status, using an overlap weight matching strategy. Patients will be matched on age, gender, ethnicity, Elixhauser comorbidity index and month of admission as well as severity of acute illness (need for intensive care unit and acute organ failure score present-on-admission), performance of rapid diagnostic testing for bacterial respiratory pathogens, and receipt of concomitant putative COVID-19 directed therapy (remdesivir, tocilizumab, systemic corticosteroids, hydroxychloroquine) initiated on the day of or day after admission respectively. Logistic regression will be performed downstream to matching to mitigate the impact of residual confounding.The primary outcome and secondary outcomes are reported separately below.

Effect modification of the relationship between empiric antibiotics and outcomes will be examined across clinically relevant subgroups based on antibiotic regimens (separately comparing community and hospital acquired type coverage to no empiric antibiotics respectively), and those with or without need for non-invasive ventilation on admission as well as quartiles of hospital's frequency of empiric antibiotic use and admission procalcitonin level (when available) respectively among patients admitted with COVID-19.

Sensitivity analyses will be performed to examine outcomes with vs without coding for conditions that may or may not suggest a definite indication for antibiotic on admission (e.g. chronic obstructive lung disease exacerbation) and/or explicit diagnosis for "sepsis" (as it remains unclear in whom this code was indicated to represent confirmed viral sepsis). Sensitivity analyses will also be performed to include patients without diagnosis codes for acute lower respiratory illness present-on-admission to include patients with COVID-19 pneumonia who may not have been coded for pneumonia per se.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Admitted to hospital with International Classification of Diseases Version 10 (ICD-10) diagnosis coding COVID-19 present-on-admission or positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) polymerase chain reaction test sampled on admission
* Patients admitted to hospital with ICD-10 diagnosis coding for pneumonia present-on-admission

Exclusion Criteria:

* Patients with suspected extra-pulmonary bacterial infection
* Patients receiving mechanical ventilation or vasopressors within 48 hours of arrival
* Patients coded as having septic shock present on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients admitted to hospital with a diagnosis of COVID-19 on arrival as defined by ICD-10 code or legacy coding for coronavirus (prior to implementation of new ICD-10 code) and/or a positive SARS-CoV-2 polymerase chain reaction test on admission. Patients included will have no other sources of infection identified on admission and will be clinically stable.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
In-Hospital Mortality or discharge to hospice | From time of admission to death during the hospitalization or discharge to hospice
  Death during the hospitalization or discharge to hospice

SECONDARY OUTCOMES:
Rates of Mechanical Ventilation | From 48 hours post admission to discharge or death
  Mechanical ventilation initiated after 48 hours into the admission as a marker of clinical deterioration and its relationship to receipt of empiric antibiotic
Rates of C. difficile infection | not present-on-admission
  Identify the risk of C. difficile infection on patients according to empiric therapy status as captured by diagnosis codes not present-on-admission
Length of stay for survivors | From admission to discharge (not to hospice)
  As a marker of morbidity and and its relationship to receipt of empiric antibiotic therapy
Rates of ICU Admission | From 48 hours post admission to discharge
  As a marker of clinical deterioration and its relationship to receipt of empiric antibiotic therapy among patients who did not require ICU admission upon arrival
Rates of Acute Kidney Injury | not present-on-admission
  Identify the risk of acute kidney injury according to empiric therapy status as captured by diagnosis codes not present-on-admission
Days free of antibiotics | 5 days from admission to discharge or primary outcome
  For patients in hospital for at least 5 days
Rates of secondary infections due to antibiotic resistant pathogens | not present-on-admission
  As above, as captured by diagnosis codes not present-on-admission

CONTACTS AND LOCATIONS:
Overall Officials: Sameer S Kadri, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No